CLINICAL TRIAL: NCT01683773
Title: A Phase I, Open Label Trial to Evaluate the Safety and Immunogenicity of AERAS-402 Followed by MVA85A in BCG Vaccinated Adults (TB032)
Brief Title: Safety Study of Tuberculosis Vaccines AERAS-402 and MVA85A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Aeras (Other); Crucell Holland BV (Industry); Emergent BioSolutions (Industry); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB032
Record Dates: First submitted 2012-08-24; First posted 2012-09-12 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Phase I; MVA85A; AERAS-402
MeSH Terms: conditions — Tuberculosis | interventions — AERAS-402; MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Two doses of AERAS-402 (1x10^11 vp intramuscular injection) followed by one dose of MVA85A (1x10^8 pfu intradermal injection)
  Interventions: Biological: AERAS-402; Biological: MVA85A
- Group B (Experimental): One dose of AERAS-402 (1x10^11 vp intramuscular injection) followed by one dose of MVA85A (1x10^8 pfu intradermal injection)
  Interventions: Biological: AERAS-402; Biological: MVA85A
- Group C (Experimental): Three doses of AERAS-402 (1x10^11 vp intramuscular injection)
  Interventions: Biological: AERAS-402

INTERVENTIONS:
Biological: AERAS-402 — Intramuscular needle injection 1x10^11 vp
  Other Names: Ad35 TB-S
Biological: MVA85A — Intradermal needle injection 1x10^8 pfu
  Other Names: AERAS-485
  Arms: Group A; Group B

SUMMARY:
This trial will investigate the administration of two new tuberculosis vaccines, called AERAS-402 and MVA85A. The purpose of this trial is to assess what happens when both of these vaccines are given one after the other. The trial will assess the safety of both vaccines and also their ability to stimulate an immune response within the body. It is hoped that when these two vaccines are given in sequence, the combined immune response is even better than when each vaccine is used individually.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the trial:

* Healthy adult aged 18-55 years
* Resident in or near Oxford (for CCVTM) or Birmingham (for WTCRF; and able to travel to Oxford for vaccinations) for the duration of the trial period
* No relevant findings in medical history or on physical examination
* Confirmation of prior vaccination with BCG not less than 6 months prior to projected trial vaccination date (by visible BCG scar on examination or written documentation)
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception for the duration of the trial period (females only)
* Refrain from blood donation during the trial
* Give written informed consent
* Allow the Investigator to register subject details with a confidential database to prevent concurrent entry into clinical trials
* Agrees to avoid elective surgery for the duration of the trial
* Has a body mass index (BMI) between 18 and 33 (weight/height2) by nomogram
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements

Exclusion Criteria:

Subjects must meet none of the following criteria to enter the trial:

* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Shared a residence within one year prior to day 0 with an individual on anti-tuberculosis treatment or with culture- or smear-positive pulmonary tuberculosis
* Previous treatment for active or latent tuberculosis infection
* Received a TST within 90 days prior to day 0
* Received a systemic antibiotic within 14 days prior to day 0
* Inability to discontinue daily medications other than the following during the trial: oral contraceptives, vitamins, nonprescription nutritional supplements, aspirin, antihistamines, antihypertensives, antidepressants, inhaled steroids, bronchodilators, and any other stable, regular medication not deemed to have an impact on safety or immunogenicity.
* Previous vaccination with candidate vaccine MVA85A or candidate vaccine FP85A or any other recombinant MVA or adenoviral vaccine; AERAS-402; or any other investigational M. tb vaccine
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), autoimmune disease, cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine, including eggs
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the subject in the triala
* Positive HBsAg, HCV or HIV antibodies
* Female currently lactating, confirmed pregnancy or intention to become pregnant during trial period
* Use of an investigational medicinal product or non-registered drug, live vaccine, or medical device other than the trial vaccine for 30 days prior to dosing with the trial vaccine, or planned use during the trial period
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned trial vaccination date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the subject at risk or may influence the result of the trial or may affect the subject's ability to participate in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety of AERAS-402 followed by MVA85A | 3 months after final vaccination
  To evaluate the safety profile of multiple doses of AERAS-402 alone, compared to one and two doses of AERAS-402 followed by MVA85A in healthy, BCG vaccinated adults, measured by number and severity of local and systemic adverse events

SECONDARY OUTCOMES:
Immunogenicity of AERAS-402 followed by MVA85A | 12-18 months after first vaccination
  To evaluate and compare the immune responses as described by flow cytometric intracellular cytokine staining, antibody serology, and Elispot assays of multiple doses of AERAS-402 alone, compared to one and two doses of AERAS-402 followed by MVA85A in healthy, BCG vaccinated adults

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital, Oxford, Oxfordshire
  - The Wellcome Trust Clinical Research Facility (WTCRF), University of Birmingham, Birmingham, West Midlands

REFERENCES:
- [Derived] Sheehan S, Harris SA, Satti I, Hokey DA, Dheenadhayalan V, Stockdale L, Manjaly Thomas ZR, Minhinnick A, Wilkie M, Vermaak S, Meyer J, O'Shea MK, Pau MG, Versteege I, Douoguih M, Hendriks J, Sadoff J, Landry B, Moss P, McShane H. A Phase I, Open-Label Trial, Evaluating the Safety and Immunogenicity of Candidate Tuberculosis Vaccines AERAS-402 and MVA85A, Administered by Prime-Boost Regime in BCG-Vaccinated Healthy Adults. PLoS One. 2015 Nov 3;10(11):e0141687. doi: 10.1371/journal.pone.0141687. eCollection 2015. PMID 26529238
- See also: The Jenner Institute - Clinical Trials — http://www.jenner.ac.uk/clinicaltrials